CLINICAL TRIAL: NCT04506398
Title: Translational Study of Molecular-subtype Heterogeneity and Evolution Pattern in Patients With hepatoceLlular Carcinoma Post-transplant Relapse - HELP 2020 Cohort Study
Brief Title: Heterogeneity and Evolution of hepatoceLlular Carcinoma in Post-transplant HCC Recurrence
Acronym: HELP-2020
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Renji-IIT-2020-0007
Record Dates: First submitted 2020-08-06; First posted 2020-08-10 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Hepatocellular Carcinoma Recurrent; Liver Transplant; Complications
MeSH Terms: interventions — Liver Transplantation; Exome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective cohort: 20 HCC patients experienced post-transplant HCC
  Interventions: Procedure: liver transplant; Diagnostic Test: whole exome sequencing
- Perspective cohort: 20 HCC patients who underwent liver transplant, the patients would be recruited if recurrence would be diagnosed >6 months after liver transplant
  Interventions: Procedure: liver transplant; Diagnostic Test: ctDNA; Diagnostic Test: whole exome sequencing

INTERVENTIONS:
Procedure: liver transplant — Liver transplantation for hepatocellular carcinoma has the potential to eliminate both the tumor as well as the underlying cirrhosis and is the ideal treatment for HCC in cirrhotic liver as well as massive HCC in noncirrhotic liver.
Diagnostic Test: ctDNA — Circulating Tumor DNA Correlates With Microvascular Invasion and Predicts Tumor Recurrence of Hepatocellular Carcinoma
  Groups: Perspective cohort
Diagnostic Test: whole exome sequencing — xome sequencing analysis of liver tumors could reveal mutational signatures associated with specific risk factors of recurrence.

SUMMARY:
Objective of Study: This study will evaluate the heterogeneity and evolution pathway between primary HCC and tumor relapse after liver transplant.

According to the "Seed-Soil" theory, the primary hypothesis of this study is that HCC patients with different molecular-subtype experience altered different pattern of post-transplant recurrence, thus may have altered postoperative Recurrence-Free Survival (RFS). Because the donors' liver construct different microenvironment for CTC(circulating tumor cells) colonization. The investigators design this translational study to ①explore potential high recurrent risk HCC molecular-subtypes which might benefit from neoadjuvant systematic therapy or early adjuvant systematic therapy;②identify the molecular subtype heterogeneity of primary and recurrent HCC to guide the precision medicine.

DETAILED DESCRIPTION:
40 specimens will be obtained from the primary tumor during liver transplant surgery and biopsy/specimens from intrahepatic tumor or lung metastasis when the patients experience postoperative relapse. The molecular-subtype of HCC will be determined via whole exom sequence(WES), immunohistochemistry(IHC) and RNA-Seq.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically or cytologically or by radiological criteria proven hepatocellular carcinoma; known mixed histology (e.g. hepatocellular carcinoma plus cholangiocarcinoma) or fibrolamellar variant is not allowed
* Patients have post-transplant HCC recurrence(cohort 1), Indication for being an candidate in the waiting list for liver transplant according to multidisciplinary board evaluation(cohort 2)
* The time frame between liver transplant and diagnosis of post-transplant HCC recurrence> 6 months
* No prior hepatectomy or systemic therapy or local therapy (TACE etc.)

Exclusion Criteria:

* History of oncological systemic treatment
* early recurrence(<6 months)
* multiple organ transplantation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort 1: HCC patients experienced post-transplant HCC Cohort 2: High recurrence-risk HCC patients who underwent liver transplant
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-09-10 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
molecular-subtype heterogeneity between primary HCC and post-transplant HCC recurrence | up to 2 years
  It is defined as the change of HCC molecular subtype by comparing the primary tumor with intrahepatic or intrapulmonary recurrent tumor.

SECONDARY OUTCOMES:
molecular-subtype | up to 2 years
  I.Progenitor Type: defined by the transcriptional and protein overexpression of hepatic progenitor markers, inactivating mutations in RPS6KA3 and AXIN1 and hyperphosphorylation of ERK. The main signalling pathways specifically activated in the progenitor subclass are IGF1R and AKT.
  II.TGFβ-Wnt Type: characterised by activation of both TGFβ and Wnt pathways and an exhausted immune response. Also, an enrichment in TP53 inactivating mutations, amplification of FGF19 and CCND1, as well as frequent activation of pro-survival signalling pathways including cell cycle, mTOR, RAS-MAPK and MET can be detected.
  III.G4 Type: It frequently harbour a steatohepatitic phenotype, as well as exhibiting activation of the IL6/JAK-STAT pathway.
  IV.CTNNB1 Type: a subset of HCC harbouring CTNNB1 mutations. TERT promoter mutations are more frequent in this subclass
Recurrence-Free Survival (RFS) | up to 3 years
  RFS is defined as the time from inclusion to first documentation of disease recurrence (intrahepatic or intrapulmonary) as assessed by BICR or by pathology consistent with HCC if required per the site's standard of care, or death due to any cause (both cancer and non-cancer causes of death)

CONTACTS AND LOCATIONS:
Overall Officials: Hao Feng, M.D., Ph.D., Study Director — Dept. of Liver surgery, Renji Hospital, Medical School of Shanghai Jiaotong University
Locations (1):
- Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, China